CLINICAL TRIAL: NCT07382193
Title: Evaluation of the Eight - Strand Repair of Flexor Tendon Injuries Without Splinting a Prospective Cohort Study
Brief Title: Evaluation of Eight-Strand Flexor Tendon Repair Without Splinting
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdalrhaman Mohamed Nasr Eldin Mohamed, Resident at Orthopaedics and Traumatology Department, Assiut University, Assiut University
Other Study IDs: Eight-strand Tendon Repair
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Flexor Tendon Injury; Splints; Flexor Tendon Repair; Flexor Tendon
Keywords: Eight-strand repair; Flexor tendon injury; no splint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This prospective cohort study evaluates functional outcomes of primary eight-strand flexor tendon repair in zone II without postoperative splinting in 40 adults (≥18 years) at Assiut University Hospitals. Patients undergo wide-awake local anesthesia no tourniquet (WALANT) surgery followed by immediate gentle active motion. Primary outcome: total active motion via Strickland score at 6 weeks and 6 months. Secondary: grip strength, DASH score, patient satisfaction.

DETAILED DESCRIPTION:
Flexor tendon injuries in zone II are traditionally managed with postoperative splinting to protect the repair, but this can limit early mobilization and functional recovery. This prospective cohort study aims to evaluate the clinical and functional outcomes of primary flexor tendon repair using an eight-strand core suture technique without postoperative splinting.

All procedures will be performed under wide-awake local anesthesia without a tourniquet (WALANT). The injured tendons will be repaired using an innovative crossed eight-strand core suture technique with PDS 3-0 or 4-0 sutures, depending on tendon size. Standard aseptic technique and microsurgical instruments will be utilized.

Unlike traditional protocols, no splint will be applied postoperatively. Patients will begin gentle, active range-of-motion exercises starting on postoperative day 5. This approach aims to leverage the superior tensile strength of the eight-strand repair to allow early mobilization, potentially reducing adhesion formation and improving outcomes.

Patients will be followed up weekly until 6 weeks, then at 12 weeks, and finally at 6 months post-surgery. Skin sutures will be removed at two weeks.

The primary outcome is Total Active Motion (TAM) assessed using the Strickland and Glogovac score at 6 weeks and 6 months. Secondary outcomes include grip strength and patient-reported function via the Disability of the Arm, Shoulder, and Hand (DASH) questionnaire at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+ years).
* Single or multiple clean-cut flexor tendon injuries.
* Primary repair performed within 2 weeks.
* Patients with concurrent digital nerve injuries will include if the nerve could be directly repaired.

Exclusion Criteria:

* Crush or avulsion injuries.
* Associated fractures or neurovascular compromise.
* Recurrent or chronic tendon injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) presenting to Assiut University Hospitals with single or multiple clean-cut flexor tendon injuries in zone II, eligible for primary repair within 2 weeks of injury. Concurrent directly repairable digital nerve injuries are included. Crush/avulsion injuries, associated fractures, neurovascular compromise, or recurrent/chronic cases are excluded. Target enrollment: 40 patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Total Active Motion (Strickland Score) | 6 weeks and 6 months post-surgery
  Total active motion of the injured finger(s) measured using the Strickland and Glogovac score via handheld goniometer, assessing flexion excursion.

SECONDARY OUTCOMES:
Grip Strength | 6 weeks and 6 months post-surgery
  Grip strength of the injured hand measured using a standard hand dynamometer.